CLINICAL TRIAL: NCT01024322
Title: Collagen Crosslinking With Ultraviolet-A in Asymmetric Corneas
Status: Terminated | Type: Observational
Why Stopped: Terminated to initiate FDA IND-cleared study protocol
Sponsor: Cxlusa (Industry)
Responsible Party: Sponsor
Other Study IDs: CXL
Record Dates: First submitted 2009-10-28; First posted 2009-12-02 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-09

CONDITIONS: Keratoconus; Ectasia; Degeneration
Keywords: Diagnosis of keratoconus, post-LASIK ectasia, FFKC, or pellucid marginal degeneration
MeSH Terms: conditions — Keratoconus; Dilatation, Pathologic | interventions — Moxifloxacin; Ketorolac Tromethamine; Steroids; Fluorometholone; prednisolone acetate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Ciprofloxicine or Vigamox or other.
  Interventions: Drug: Ciprofloxicine or Vigamox or other.
- Nonsteroidal (Acular, Voltaren Xibrom, etc)
  Interventions: Drug: Nonsteroidal (Acular, Voltaren Xibrom, etc)
- Steroid (FML, Pred Forte, Flarex, etc.)
  Interventions: Drug: Steroid (FML, Pred Forte, Flarex, etc.)

INTERVENTIONS:
Drug: Ciprofloxicine or Vigamox or other. — Ciprofloxicine or Vigamox or other to be used qid till epithelialized.
  Groups: Ciprofloxicine or Vigamox or other.
Drug: Nonsteroidal (Acular, Voltaren Xibrom, etc) — Nonsteroidal (Acular, Voltaren Xibrom, etc) used up to qid for up to 5-10 days post-op
  Groups: Nonsteroidal (Acular, Voltaren Xibrom, etc)
Drug: Steroid (FML, Pred Forte, Flarex, etc.) — Steroid (FML, Pred Forte, Flarex, etc.) to be used qid for 8 weeks.
  Groups: Steroid (FML, Pred Forte, Flarex, etc.)

SUMMARY:
To evaluate the efficacy of ultraviolet-A (UVA)-induced cross-linking of corneal collagen (CXL) as a method to increase the biomechanical and biochemical stability of the cornea by inducing additional cross-links within or between collagen fibers using UVA light and the photo- mediator riboflavin. The purpose of this study is to generate data for presentation at medical meetings and for peer-review publication

ELIGIBILITY:
Inclusion Criteria:

* 8 years of age or older
* Diagnosis of keratoconus, post-LASIK ectasia, or pellucid marginal degeneration or forme fruste pellucid marginal degeneration.
* Diagnosis of FFKC
* History of Radial Keratotomy with fluctuating vision.
* Terrien's Marginal Degeneration
* Ability to provide written informed consent
* Likely to complete all study visits
* Minimum corneal thickness of at least 300 250 microns measured by ultrasound or Pentacam for all indications other than Terriens. For Terriens, the minimal corneal thickness should be consistent with the surgeon's best surgical judgment.

Exclusion Criteria:

* Severe corneal scarring that markedly affects vision
* Contraindications to any study medications or their components
* Pregnancy or breast feeding
* Active Herpes Corneal Disease

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinic.
Sampling Method: Probability Sample
Enrollment: 1189 (Actual)
Dates: Start 2009-10-01 (Actual); Primary Completion 2017-02-03 (Actual); Study Completion 2017-02-03 (Actual)

PRIMARY OUTCOMES:
Increase the biomechanical and biochemical stability of the cornea by inducing additional cross-links within | 1 year

SECONDARY OUTCOMES:
increase the biomechanical and biochemical stability of the cornea between collagen fibers using UVA light and the photo- mediator riboflavin | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: William Trattler, MD, Principal Investigator — The Center for Excellence in Eye Care; Roy Rubinfeld, MD, Principal Investigator — Re: Vision
Locations (3):
- United States (3):
  - The Center for Excellence in Eye Care, Miami, Florida
  - TLC Laser Eye Center, Rockville, Maryland
  - TLC Laser Eye Center, Fairfax, Virginia